CLINICAL TRIAL: NCT05229887
Title: Confirmation of Tube Placement in Newborns
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: need to be redesigned
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00116201
Record Dates: First submitted 2022-01-31; First posted 2022-02-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-04

CONDITIONS: Respiratory Distress Syndrome; Apnea of Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nostril-Tragus-Length (Active Comparator)
  Interventions: Procedure: Nostril-Tragus-Length
- Vocal cord markings (Experimental)
  Interventions: Procedure: Vocal cord marking

INTERVENTIONS:
Procedure: Nostril-Tragus-Length — Endotracheal tube depth is determined by measuring the newborn's nasal septum-tragus length (NTL) and adding 1cm.
  The NTL is described as the distance from the base of the nasal septum to the tragus of the ear.
  Arms: Nostril-Tragus-Length
Procedure: Vocal cord marking — The endotracheal tube has markings on the tube, which are called vocal cord markings, which will be used to provide a guidance to how deep to place the ETT into the trachea.
  Arms: Vocal cord markings

SUMMARY:
Tracheal intubation remains a common procedure in the neonatal intensive care unit (NICU) and the delivery room (DR).

Current guidelines recommend Estimation of correct endotracheal tube (ETT) insertion Our hospital policy recommends to estimate the correct depth (cm) of tube placement by measuring the nasal-ear-tragus length using the "7-8-9 rule" when the endotracheal tube is placed orally. Using this formula an infant weighing 1kg would be intubated to a depth of 7cm, a 2kg infant to a depth of 8cm, and a 3kg infant to a depth of 9cm from the upper lip.

With the new 2015 guidelines, ETT depth is determined by measuring the newborn's nasal septum-tragus length (NTL) and adding 1cm or by using the "initial endotracheal tube insertion depth" table. The NTL is described as the distance from the base of the nasal septum to the tragus of the ear.

However, studies using NTL reported that using this technique only resulted in correct ETT placement in 56% of cases.

Every ETT has markings on the tube, which are called vocal cord markings, which are to be used to provide a guidance to how deep to place the ETT into the trachea. There has been npc study to compare the vocal cord markings with the current approach of NTL.

The current study aims to determine if the use of vocal cord markings during intubation increases percentage of correct endotracheal tube placement compared to NTL in preterm and term infants.

ELIGIBILITY:
Inclusion Criteria:

* All infants (term and preterm) born at The Royal Alexandra Hospital who require endotracheal intubation in the delivery room or/and Neonatal Intensive Care Unit will be eligible.

Exclusion Criteria:

* Infants will be excluded if their parents refuse to give consent to this study.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of endotracheal tubes correctly placed within the trachea | within 30 minutes after endotracheal intubation

SECONDARY OUTCOMES:
Mortality in the Neonatal Intensive Care Unit | 0-200 days
  We will record the number of infants who die during their admission
Necrotizing Enterocolitis | 0-200 days
  We will record the number of infants who are diagnosed with Necrotizing Enterocolitis
Patent Ductus Arteriosus | 0-200 days
  We will record the number of infants who are diagnosed with Patent Ductus Arteriosus
Intraventricular hemorrhage all grades | 0-200 days
  We will record the number of infants who are diagnosed with intraventricular hemorrhage
Bronchopulmonary Dysplasia at | 36 weeks corrected gestational age
  We will record the number of infants who are diagnosed with Bronchopulmonary Dysplasia
Changes in oxygen saturation during intubation procedure | 0 to 60 seconds
  During intubation we will record the lowest oxygen saturation
Changes in Heart rate during intubation procedure | 0 to 60 seconds
  During intubation we will record the lowest heart rate.
Duration of Intubation procedure | 0 to 60 seconds
  During Intubation, we will measure time from end of mask ventilation to connection of the ventilation device to ETT
Airway injury observed during intubation (including blood, swollen cords, vocal cord redness) | 0 to 60 seconds
  Observed by the person who performs the intubation by looking for blood, swollen cords, redness. There is no score or questionnaire. The operator will only assess these with yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Investigators can contact the PI to discuss to use the collected data
Supporting Information: Study Protocol, ICF, CSR